CLINICAL TRIAL: NCT04552522
Title: Immunological Response After Shrimp Oral Immunotherapy Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 090/2563
Record Dates: First submitted 2020-09-13; First posted 2020-09-17 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Allergy to Shrimp; Immunotherapy
Keywords: Shrimp allergy; Oral immunotherapy; Specific Immunoglobulin E; Skin sensitization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Shrimp allergy with Intend to eat shrimp (Experimental): Case shrimp Immunoglobulin E mediated allergy and intend to eat shrimp and start oral immunotherapy for shrimp
  Interventions: Other: shrimp allergy with intend to eat shrimp
- Shrimp allergy with avoid shrimp (No Intervention): Case shrimp allergy with avoid shrimp

INTERVENTIONS:
Other: shrimp allergy with intend to eat shrimp — shrimp allergy with intend to eat shrimp and treat with oral immunotherapy
  Arms: Shrimp allergy with Intend to eat shrimp

SUMMARY:
Oral immunotherapy is effective in desensitized food allergy. Shrimp allergy is increasing in Thailand. So the purpose of our study is to determine level of specific immunoglobulin E antibodies to shrimp, Immunoglobulin G4 and immunoblot analysis in shrimp allergy patients after shrimp oral immunotherapy.

DETAILED DESCRIPTION:
All subject in this study were sensitized to shrimp. All patient was clinically evaluated, with focus on shrimp allergy by medical history, medical examination and gold standard oral food challenge test. Compare oral immunotherapy to shrimp and shrimp avoidance. Blood sample was taken for baseline determination of immunoglobulin E antibodies to shrimp. The primary outcome was the specific immunoglobulin E antibodies to shrimp,Immunoglobulin G4 and immunoblot analysis in case that oral immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 12 - 40 years old
* History of Immunoglobulin E-mediated shrimp allergy > 3 episode/year or disturb quality of life
* Positive oral food challenge test for shrimp

Exclusion Criteria:

* History of shrimp anaphylaxis (include cardiovascular or neurological symptoms)
* Shellfish dependent exercise induced anaphylaxis
* History of cardiovascular disease, uncontrolled asthma, severe atopic dermatitis
* History of Beta-blocker, Angiotensin-converting enzyme inhibitor, Angiotensin receptor blocker, Calcium channel blocker

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
specific Immunoglobulin E, Immunoglobulin G4, immunoblot analysis from Desensitized to shrimp allergen | 1 year
  To follow-up the level of specific Immunoglobulin E, Immunoglobulin G4, immunoblot analysis from Desensitized to shrimp allergen

SECONDARY OUTCOMES:
Adverse event from Shrimp oral immunotherapy | 1 year
  To follow up adverse event from Shrimp oral immunotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Punchama Pacharn, MD, Principal Investigator — Mahidol University
Locations (1):
- Siriraj Hospital, Bangkoknoi, Bangkok, Thailand

REFERENCES:
- [Background] Pajno GB, Fernandez-Rivas M, Arasi S, Roberts G, Akdis CA, Alvaro-Lozano M, Beyer K, Bindslev-Jensen C, Burks W, Ebisawa M, Eigenmann P, Knol E, Nadeau KC, Poulsen LK, van Ree R, Santos AF, du Toit G, Dhami S, Nurmatov U, Boloh Y, Makela M, O'Mahony L, Papadopoulos N, Sackesen C, Agache I, Angier E, Halken S, Jutel M, Lau S, Pfaar O, Ryan D, Sturm G, Varga EM, van Wijk RG, Sheikh A, Muraro A; EAACI Allergen Immunotherapy Guidelines Group. EAACI Guidelines on allergen immunotherapy: IgE-mediated food allergy. Allergy. 2018 Apr;73(4):799-815. doi: 10.1111/all.13319. Epub 2017 Dec 5. PMID 29205393